CLINICAL TRIAL: NCT01582152
Title: Phase I/II Adaptive Randomized Trial of Bevacizumab Versus Bevacizumab Plus TPI 287 in Adults With Recurrent Glioblastoma
Brief Title: Phase I/II Bevacizumab Versus Bevacizumab Plus TPI 287 for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 2 part of the trial will no longer continue since the protocol competes with another TPI287 protocol in outside institution supported by the sponsor.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0705; NCI-2012-00846 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Brain Neoplasms; Central Nervous System Neoplasms
Keywords: Brain Neoplasms; Central Nervous System Neoplasms; Recurrent Glioblastoma; Glioblastoma multiforme; GBM; Gliosarcoma; TPI287; Bevacizumab; Avastin; Anti-VEGF Monoclonal Antibody; rhuMAb-VEGF
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — TPI-287; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TPI 287 + Bevacizumab (Experimental): Part I: Patients assigned to receive 1 of 4 dose levels of TPI 287 based on when joining the study.
  Phase I Starting Dose of TPI287 160 mg/m2 given by vein on Day 1 every three weeks of a 42 Day cycle. Bevacizumab given at 10 mg/kg by vein on Day 1 every 2 weeks of a 42 Day cycle.
  Phase II Starting Dose of TPI287: Maximum Tolerated Dose (MTD) from Phase I.
  Interventions: Drug: TPI287; Drug: Bevacizumab
- Bevacizumab Group (Experimental): Phase II: Participants randomized to Arm A (bevacizumab alone at 10 mg/kg every 2 weeks) versus Arm B (bevacizumab at 10 mg/kg every 2 weeks plus TPI 287.
  Participant may enroll in Crossover Group to receive TPI 287 and bevacizumab if disease gets worse at any time during treatment with bevacizumab alone.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: TPI287 — Phase I Starting Dose: 160 mg/m2 given by vein on Day 1 every three weeks of a 42 Day cycle.
  Phase II Starting Dose: Maximum Tolerated Dose (MTD) from Phase I.
  Arms: TPI 287 + Bevacizumab
Drug: Bevacizumab — Arm A + B: 10 mg/kg by vein every 2 weeks of a 42 day cycle.
  Other Names: Avastin; Anti-VEGF Monoclonal Antibody; rhuMAb-VEGF

SUMMARY:
The goal of Part I of this clinical research study is to find the highest tolerable dose of TPI 287 that can be given with bevacizumab to patients with glioblastoma. The goal of Part II is to learn if TPI 287 when given with bevacizumab can help to control glioblastoma better than when bevacizumab is given alone. The safety of the drug combination will also be studied.

TPI 287 is similar to a type of chemotherapy drug called a taxane and is designed to block a protein (tubulin) that helps the cancer cells divide. By blocking the tubulin, the drug may be able to cause the cancer cells to shrink or stop growing.

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

DETAILED DESCRIPTION:
Part I and Part II of the Study:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 3 groups of 3-6 participants will be enrolled in Part I of the study. After that, up to 90 participants will be enrolled in Part II.

If you are in Part I, you will be assigned to receive 1 of 4 dose levels of TPI 287 based on when you join this study. The first 3-6 participants will receive a starting dose level. The next 3-6 participants will receive a higher dose if no intolerable side effects were seen or a lower dose if intolerable side effects were seen. Your dose may be lowered if you have side effects.

All participants will receive bevacizumab at the same dose level for the entire study.

If you are in Part II, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. If you are one of the first 20 participants in Part II, you will be randomly assigned to a group. If you are enrolled after the first 20 participants, you will be more likely to be enrolled in the group that is showing better results.

* If you are in Group 1, you will receive bevacizumab.
* If you are in Group 2, you will receive bevacizumab and TPI 287.

If the disease gets worse at any time during the treatment with bevacizumab alone, you may enroll in the Crossover Group to receive TPI 287 and bevacizumab.

Other Drugs:

If you are taking TPI 287, you will be given standard drugs such as Benadryl® (diphenhydramine) and cimetidine to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Drug Administration:

There are 42 days in each study cycle.

Part I:

* On Days 1 and 22 of every cycle, you will receive TPI 287 by vein over 1 hour.
* On Days 1, 15, and 29 of every cycle, you will receive bevacizumab by vein over 30-90 minutes.

Part II:

If you are in Group 1:

° On Days 1,15, and 29 of every cycle, you will receive bevacizumab by vein over 30-90 minutes.

If you are in Group 2 or the Crossover Group:

* On Days 1 and 22 of every cycle, you will receive TPI 287 by vein over 1 hour.
* On Days 1, 15, and 29 of every cycle, you will receive bevacizumab by vein over 30-90 minutes.

Study Visits for Part I, Group 2, or Crossover Group of Part II:

Every time you receive the study drug(s), your vital signs will be recorded before and at the end of the infusion.

On Days 1, 15, 22, and 29 of Cycle 1, blood (about 1- 2 teaspoons) will be collected for routine tests.

On Days 1, 15, and 29 of Cycle 1, urine will be collected for kidney function tests.

On Day 1 of Cycles 2 and beyond:

* Your medical history and performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have a complete physical exam, including measurement of your weight.
* You will have a neurological exam.
* Blood (about 1-2 teaspoons) will be collected for routine tests.
* Urine will be collected for kidney function tests.
* You will have an MRI scan of the brain to check the status of the disease.

On Days 15, 22, and 29 of Cycles 2 and beyond, blood (about 1-2 teaspoons) will be drawn for routine tests.

Study Visits for Group 1 of Part II:

Every time you receive the study drug(s), your vital signs will be recorded before and after the infusion.

On Days 1, 15, and 29 of Cycle 1:

* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* Urine will be collected for kidney function tests.

On Day 1 of Cycle 2 and beyond:

* Your medical history and performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have a complete physical exam, including measurement of your weight.
* You will have a neurological exam.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Urine will be collected for kidney function tests.
* You will have an MRI scan of the brain to check the status of the disease.

On Day 15 and 29 of Cycles 2 and beyond, blood (about 1-2 teaspoons) will be drawn for routine tests.

At any time during the study, extra tests may be performed if the doctor thinks they are needed for your safety. The study doctor will tell you more about any extra tests.

Length of Treatment:

You may continue taking the study drug(s) for as long as the doctor thinks it is in your best interest. If you enroll in the Crossover Group, you may continue taking the study drugs for up to 6 additional cycles in the Crossover Group.

You may no longer be able to receive the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment and follow-up visits.

End-of-Treatment Visit:

Within 28 days after you stop the study drugs:

* Your medical history and performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will have a neurological exam.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Urine will be collected for kidney function tests.
* You may have an MRI scan of the brain to check the status of the disease.

Long-Term Follow-Up:

Every 3 months after the end-of-treatment visit for up to 1 year, you will be called and asked how you are feeling. This call will take about 5-10 minutes.

This is an investigational study. TPI 287 is not FDA approved or commercially available. It is currently being used for research purposes only. Bevacizumab is FDA approved and commercially available for the treatment of brain tumors, including glioblastoma. The combination of TPI 287 and bevacizumab in glioblastoma is investigational.

Up to 108 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven glioblastoma or gliosarcoma to be eligible for this protocol. Patients will be eligible if the original histology was low-grade glioma or anaplastic glioma (WHO II or III) and a subsequent histological diagnosis of glioblastoma or gliosarcoma is made. Only patients with histologically proven or imaging proven recurrent glioblastoma or gliosarcoma will be eligible for this protocol.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan and should have failed radiation and temozolomide therapy. The scan done prior to study entry documenting progression will be reviewed by the treating physician to document changes in tumor dimension to confirm recurrence. Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis.
3. For this study, patients may have had up to 2 prior relapses provided the functional status and other eligibility criteria for enrollment are met.
4. All patients must sign an informed consent indicating their awareness of the investigational nature of this study in keeping with the policies of this hospital.
5. The baseline on-study MRI should be performed within 14 days (+/- 3 working days) prior to registration and on a steroid dosage that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and the initiation of therapy (or at that time), a new baseline MRI is required. The same type of scan, i.e., MRI, must be used throughout the period of protocol treatment for tumor measurement.
6. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: a) At least 4 weeks have elapsed from the date of surgery and the patients have recovered from the effects of surgery. b) Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study. c) To best assess the extent of residual measurable disease post-operatively, a MRI should be done no later than 96 hours in the immediate post-operative period.
7. Patients must be 18 years old or older.
8. Patients must have a Karnofsky performance status (KPS) equal or greater than 60.
9. Patients must have recovered from the toxic effects of prior therapy to < grade 2 toxicity per CTC version 4 (except deep vein thrombosis) prior to Day 1 of Cycle 1: a) at least 12 weeks from completion of radiation therapy except if there is unequivocal evidence for tumor recurrence (such as histological confirmation or advanced imaging data such as positron emission computed tomography (PET) scan in which case at least 4 weeks from completion of radiation therapy will suffice (Note: for patients who have undergone surgery to confirm recurrence after radiation therapy, guidelines in 5.2.6a should be followed). b) 4 weeks from prior cytotoxic therapy. c) 4 weeks from prior experimental drug. d) 2 weeks from vincristine.
10. 9) (continued) e) 6 weeks from nitrosoureas. f) 3 weeks from procarbazine administration. g) 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count). h) Patients who receive anticancer agents for non-therapeutic purposes unrelated to this study (such as presurgically for obtaining pharmacology data for the agent) will be eligible to enter the study provided they have recovered from the toxic effects of the agent if any. i) Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
11. Patients must have adequate bone marrow function (ANC> 1,500/mm3 and platelet count of > 100,000/mm3), adequate liver function (SGPT < 3 times upper limit normal and alkaline phosphatase < 2 times upper limit normal, total bilirubin <1.5 mg/dl), and adequate renal function (BUN and creatinine <1.5 times institutional normal) prior to starting therapy.
12. Male patients on treatment with TPI 287 must agree to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication. Women of childbearing potential must not be pregnant (as evidenced by a negative pregnancy test prior to study entry), must not be breast-feeding and must practice adequate contraception for the duration of the study, and for 30 days after the last dose of study medication. An adequate method of contraception is one highly effective method or more than one additional methods. Highly effective methods include intrauterine device (IUD), hormonal (birth control pills, injections, implants), tubal ligation and partner's vasectomy. Additional effective methods include latex condom, diaphragm and cervical cap.
13. Patient must be able to tolerate the procedures required in this study including periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study.
14. Exploratory, Cross-Over Trial Arm: Patients with evidence of clinical or radiographic progression on the bevacizumab alone arm are eligible for cross-over into the exploratory arm of the trial if KPS is 50 or greater and all other criteria for initial enrollment in the trial are still met at time of progression. Patients will be excluded if the investigators feel the patient will not tolerate TPI 287 or if an alternative treatment approach is deemed necessary by the treating physician.

Exclusion Criteria:

1. Inability to comply with protocol or study procedures.
2. Prior treatment with bevacizumab or TPI 287.
3. Patients who are receiving concurrent Enzyme-Inducing Anti-Epileptic Drugs (EIAEDs) (e.g., carbamazepine, oxcarbazepine, phenytoin, fosphenytoin, phenobarbital and primidone, or who received EIAEDs within 2 weeks prior to the first dose of study drug.
4. Patients who have received more than one course of radiation therapy or more than a total dose of 65 Gy. Patients may have received radiosurgery as part of the initial therapy (i.e., in addition to one course of radiation therapy); however, the dose used for the radiosurgery counts against the total dose limit listed above.
5. Patient who have received prior taxane chemotherapy for treatment of GBM or other malignancy. GliadelTM as part of the initial therapy is permitted. Patients who have received prior biologic therapy other than bevacizumab will be eligible.
6. Any condition, including the presence of clinically significant laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. These would include: a) Active infection including known AIDS or Hepatitis C or with a fever >/= 38.5°C within 3 days prior to the study enrollment. b) Diseases or conditions that obscure toxicity or dangerously alter drug metabolism. c) Serious intercurrent medical illness (e.g. symptomatic congestive heart failure).
7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
8. Inadequately controlled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg)
9. Prior history of hypertensive crisis or hypertensive encephalopathy
10. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
11. History of myocardial infarction or unstable angina within 6 months prior to Day 1
12. History of stroke or transient ischemic attack within 6 months prior to Day1
13. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
14. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
15. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
17. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
18. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
19. Serious, non-healing wound, active ulcer, or untreated bone fracture.
20. Proteinuria as demonstrated by: (1) Urine protein:creatinine (UPC) ratio >/= 1.0 at screening; OR (2) Urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
21. Known hypersensitivity to any component of bevacizumab
22. Pregnancy (positive pregnancy test) or lactation. Not able to use of effective means of contraception (men and women) in subjects of child-bearing potential.
23. Patients with Grade 2 or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W K Alfred Yung, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 24, 2012 to June 02, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated early without advancing to the second portion (Phase II).
Groups:
- TPI 287 160 mg/m2 + Bevacizumab: TPI287 160 mg/m2 given intravenous (IV) on Day 1 every three weeks of a 42 Day cycle. Bevacizumab given at 10 mg/kg IV on Day 1 every 2 weeks of a 42 Day cycle.
- TPI 287 140 mg/m2 + Bevacizumab: TPI287 140 mg/m2 given intravenous (IV) on Day 1 every three weeks of a 42 Day cycle. Bevacizumab given at 10 mg/kg IV on Day 1 every 2 weeks of a 42 Day cycle.
Period: Overall Study
Arm/Group | TPI 287 160 mg/m2 + Bevacizumab | TPI 287 140 mg/m2 + Bevacizumab
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Disease Progression | 4 | 5
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TPI 287 160 mg/m2 + Bevacizumab | TPI 287 140 mg/m2 + Bevacizumab | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 57.5 [35 to 72] | 52 [44 to 61] | 55 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) measured from time of registration until date of progression or death (whichever is earlier) (event time) or last date participant was known to be alive without progression (censoring time).
Time Frame: PFS will be evaluated as a continuous variable, up to one year
Measure: Median (Full Range); unit: weeks
Groups:
- TPI 287 160 mg/m2 + Bevacizumab: TPI287 160 mg/m2 IV on Day 1 every three weeks + Bevacizumab 10 mg/kg IV on Day 1 every 2 weeks of 42 Day cycle.
- TPI 287 140 mg/m2 + Bevacizumab: TPI287 140 mg/m2 IV on Day 1 every three weeks + Bevacizumab 10 mg/kg IV on Day 1 every 2 weeks of 42 Day cycle.
Arm/Group | TPI 287 160 mg/m2 + Bevacizumab | TPI 287 140 mg/m2 + Bevacizumab
Number analyzed (Participants) | 6 | 6
weeks | 12.5 [6 to 37] | 9.5 [7 to 44]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is number participants who experience complete response (CR) or partial response (PR) analyzed for completion of at least one cycle in all treatment arms, including exploratory treatment arm. CR requires: 1) complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; 2) no new lesions; 3) stable or improved non-enhancing (T2/FLAIR) lesions; 4) off corticosteroids (or on physiologic replacement doses only); 5) stable or improved clinically. Partial response (PR) requires: 1) >50% decrease compared with baseline in sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; 2) No progression of non-measurable disease; 3) No new lesions; 4) Stable or improved non-enhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; 5) corticosteroid dose at time of scan should be < dose at baseline scan; 6) Improved or stable clinically
Time Frame: 1 year
Population: Two participants, one in each arm was not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | TPI 287 160 mg/m2 + Bevacizumab | TPI 287 140 mg/m2 + Bevacizumab
Number analyzed (Participants) | 5 | 5
percentage of participants | 40 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected through 42 day treatment period.
Arm/Group | TPI 287 160 mg/m2 + Bevacizumab | TPI 287 140 mg/m2 + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 160 mg/m2 + Bevacizumab (N=6) | TPI 287 140 mg/m2 + Bevacizumab (N=6)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 160 mg/m2 + Bevacizumab (N=6) | TPI 287 140 mg/m2 + Bevacizumab (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (3) | 3 (4)
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0)
Allergic Rhinitis (Immune system disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (13) | 3 (10)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 2 (3) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bicarbonate Serum-Low (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bilirubin Changes (Investigations) | 1 (1) | 0 (0)
Bilirubin Increase (Investigations) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 2 (3)
Blurred Vision (Eye disorders) | 4 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood urea nitrogen (BUN) Increase (Investigations) | 2 (2) | 3 (5)
Chest Pain - Cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Chest Wall Pain (Cardiac disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (3)
Cholesterol High (Investigations) | 1 (1) | 1 (2)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 3 (4)
Confusion (Psychiatric disorders) | 2 (3) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
creatine phosphokinase (CPK) Increased (Investigations) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 0 (0) | 1 (2)
Cushingoid (Endocrine disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Ear And Labyrinth Disorders - (Other) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema Face (General disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 2 (3) | 1 (1)
Elevated lactate dehydrogenase (LD) (Other) (Investigations) | 2 (2) | 2 (4)
Eye Disorders - (Other) (Eye disorders) | 3 (3) | 1 (1)
Eye Infection (Eye disorders) | 1 (1) | 0 (0)
Facial Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (13) | 6 (11)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (4)
Gait Disturbance (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 5 (8)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hemoglobin Increased (Investigations) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (10) | 5 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 5 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Irritability (General disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (6) | 3 (14)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Lymphocyte Count Decreased (Infections and infestations) | 2 (11) | 5 (27)
Lymphocyte Count Increased (Infections and infestations) | 2 (7) | 0 (0)
Memory Impairment (Nervous system disorders) | 5 (9) | 4 (4)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Metabolism And Nutrition Disorders - (Other) (Metabolism and nutrition disorders) | 5 (9) | 6 (16)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle Weakness Right-Sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Neutrophil Count Decreased (Investigations) | 1 (3) | 1 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Optic Nerve Disorder (Eye disorders) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (3)
Periodontal Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 (8) | 1 (2)
Platelet Count Decreased (Investigations) | 3 (3) | 2 (2)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyramidal Tract Syndrome (Nervous system disorders) | 1 (4) | 2 (5)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 3 (3) | 5 (6)
Skin Infection (Infections and infestations) | 2 (2) | 0 (0)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 2 (3) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weight Gain (Investigations) | 0 (0) | 1 (1)
Weight Loss (Investigations) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes